CLINICAL TRIAL: NCT03349775
Title: Cardiometabolic Disease and Pulmonary Hypertension
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: After discussion with the Data Safety Monitoring Board and NIH, the randomized clinical trial involving metformin vs. placebo is terminated due to slow enrollment in the setting of the COVID-19 pandemic.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jennifer En-Sian Ho M.D., Assistant Physician in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017P001020; 1R01HL134893-01A1 (NIH)
Record Dates: First submitted 2017-06-06; First posted 2017-11-22 (Actual); Results first posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Obesity
Keywords: Pulmonary Hypertension; BMI; Echocardiography; CPET; 6-minute walk test; Cardio Metabolic disease
MeSH Terms: conditions — Obesity; Hypertension, Pulmonary | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): Metformin: 500mg twice daily for 1 week, followed by 1g twice daily for a total of 3 months.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo: 500 mgh twice daily for 1 week, followed by 1g twice daily for a total of 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — One capsule by mouth twice a day, followed by an increase to two capsules by mouth twice a day for a total of 3 months
  Arms: Metformin
Drug: Placebo — One capsule by mouth twice a day, followed by an increase to two capsules by mouth twice a day for a total of 3 months
  Arms: Placebo

SUMMARY:
This study will investigate if metformin can help people with obesity and high pressures inside their lung blood vessels. Metformin is approved by the U.S. Food and Drug Administration (FDA) to treat diabetes, but metformin is not approved by the FDA to treat pulmonary hypertension.

This study will examine whether Metformin will improve the high pressure inside lung blood vessels in people who are obese. The study will help understand the effect of metformin on pressures inside lung blood vessels.

DETAILED DESCRIPTION:
Obesity can predispose people to develop high pressures inside their lung blood vessels, a condition called pulmonary hypertension, Pulmonary hypertension in turn, can lead to shortness of breath and other health complications such as heart failure. In this study, we seek to identify individuals at risk for the development of high pressures inside lung vessels based on BMI and dyspnea grade 1.

Participants will be screened by echocardiography to estimate pulmonary pressures. Potential participants will undergo invasive cardiopulmonary exercise testing with hemodynamic monitoring, in order to identify individuals with abnormal pulmonary vascular function either at rest or during exercise. Patients who have undergone clinically-indicated cardiopulmonary exercise testing and meet inclusion/exclusion criteria will also be recruited. Those with abnormal pulmonary vascular function will be randomized to receive Metformin or placebo for a total of 3 months under an IND exemption. The primary outcomes include the effect on pulmonary vascular function at rest and during exercise. Secondary outcomes include change in pulmonary artery endothelial cell phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years
* History of obesity and current BMI ≥ 25 kg/ m2 for study volunteers or BMI ≥ 25 kg/ m2 for those with clinically indicated CPET or known HFpEF
* History of Dyspnea (Grade 1 or more)
* Able to provide informed consent and willing to comply with study

Exclusion Criteria:

* History of diabetes mellitus
* History of primary pulmonary arterial hypertension
* History of moderate to severe COPD
* History of severe Obstructive Sleep apnea
* History of renal disease (eGFR< 45 mL/min/1.732)
* History of severe liver disease
* History of cardiovascular disease (recent heart attack or stroke) except known HFpEF
* History of blood clot in lung
* History of Splenectomy
* History of Active Cancer
* Platelets count of < 75,000
* International normalized ration (INR) of > 1.5
* History of recent anemia (HB < 9g/dL)
* Current use of Metformin
* Prior LVEF < 50% on echocardiogram
* Indication of severe valvular disease on echo
* Pregnant or planning to become pregnant in next 4 months
* History of HIV infection

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Ho, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin: 500mg tablet orally twice daily for 1 week, followed by two 500mg tablets orally twice daily for a total of 3 months.
- Placebo: Placebo: 500 mg tablet orally twice daily for 1 week, followed by two 500 mg tablets orally twice daily for a total of 3 months.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 10 | 11
Completed | 8 | 7
Not Completed | 2 | 4
Not completed — Side Effects | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — No primary outcome measurements | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population includes participants who completed the assigned arm (metformin or placebo) and were included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 60 (10) | 63 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: inches] | 65.1 (2.9) | 67.7 (4.2) | 66.3 (3.7)
Weight [Mean (Standard Deviation); unit: pounds] | 212.9 (44.1) | 224.0 (32.9) | 218.1 (38.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.3 (6.0) | 34.4 (4.6) | 34.9 (5.2)
Heart Rate (HR) [Mean (Standard Deviation); unit: beats per minute (bpm)] | 70 (13) | 70 (15) | 70 (14)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 133 (18) | 142 (14) | 137 (17)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 80 (8) | 86 (11) | 83 (9)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Vascular Hemodynamics (Rest)
Description: The metformin and placebo groups will be compared with respect to resting mean pulmonary artery pressure (mmHg)
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 8 | 7
mmHg | -3.00 (5.35) | -0.43 (4.89)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.35, t-test, 2 sided; Median Difference (Final Values) = -2.57, 95% CI 2-sided [-8.32 to 3.18], Standard Deviation 5.14

2. Primary Outcome: Pulmonary Vascular Hemodynamics (Exercise)
Description: The metformin and placebo groups will be compared with respect to augmentation of mean pulmonary artery pressure divided by augmentation of cardiac output during cardiopulmonary exercise testing (change in mean PAP divided by change in cardiac output from rest to peak exercise)
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mmHg/L/min
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 8 | 7
mmHg/L/min | -0.29 (0.83) | -1.42 (3.00)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.37, t-test, 2 sided; Median Difference (Final Values) = 1.13, 95% CI 2-sided [-1.65 to 3.92], Standard Deviation 2.13

3. Secondary Outcome: Effect on Pulmonary Artery Endothelial Cell Phenotypes
Description: We will compare the metformin and placebo groups. Specifically we will examine the following pulmonary artery endothelial cell phenotypes:
  (1) activation of phospho-eNOS as detected by immunofluorescence staining
Time Frame: baseline and 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the metformin and placebo groups over the course of the 3 months on randomized assignment to study drug.
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 8/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=10) | Placebo (N=11)
Left arm numbness and chest pain (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=10) | Placebo (N=11)
Acid Reflux (Gastrointestinal disorders) | 1 (2) | 0
GI upset (e.g. nausea, diarrhea, vomiting, abdominal discomfort, flatulence) (Gastrointestinal disorders) | 7 (11) | 4 (5)
Fatigue/Weakness (General disorders) | 0 | 2
Itching and rash/hives (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Muscle or joint soreness (Musculoskeletal and connective tissue disorders) | 0 | 3
Asthma Flare (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-Specific Symptoms (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
After discussion with the Data Safety Monitoring Board and NIH, the randomized clinical trial involving metformin vs. placebo was terminated due to slow enrollment in the setting of the COVID-19 pandemic, resulting in small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03349775/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT03349775/SAP_001.pdf
  • Informed Consent Form (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03349775/ICF_002.pdf